CLINICAL TRIAL: NCT04407338
Title: Study of the Efficacy and Tolerance of the B-Dyn Medical Device Compared to a Conventional Bolted Fusion With or Without Cage in the Treatment of Degenerative Lumbar Stenosis, With or Without Grade I Spondylolisthesis on the Degree of Postoperative Functional Disability, Preservation of Mobility and Prevention of the Adjacent Syndrome". Interventional, Prospective, Comparative, Randomized, Non-inferiority, Single Blind, International, Multicenter Clinical Study
Brief Title: Efficacy and Tolerance Study of B-DYN Versus Conventional Fusion in the Treatment of Lumbar Stenosis on the Degree of Post-operative Functional Incapacity (BDYNCLIN)
Acronym: BDYNCLIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Medical (Industry)
Collaborators: Cousin Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3001_BDYNCLIN
Record Dates: First submitted 2020-05-15; First posted 2020-05-29 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Lumbar Spinal Stenosis
Keywords: Spine; Arthrodesis; Dynamic stabilisation; BDYN
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, multicentric, comparative study of non-inferiority in parallel groups with an allocation ratio of 1:1, single-blind (the patient will be blinded from the arm of randomization), single blind (The patient will be blinded regarding randomization arm).
  The secondary objective of this study will be to assess the performance of the B-Dyn device compared to a simple fusion on dynamic parameters and the prevention of adjacent syndrome.
  Randomization, with a ratio of 1:1 will be stratified on the center and on the presence of spondylolisthesis (spondylolisthesis grade 1 on the upper instrumented (treated) level VS no spondylolisthesison the upper instrumented ( treated) level )
Who Masked: Participant
Masking Description: The patient will be blinded from the randomizing arm. As the procedure is performed under general anaesthesia, the patient will not be informed whether or not the B-Dyn® device has been implanted as a result of the procedure. The primary endpoint (the ODI being a reported outcome patient) will therefore be assessed blind to the randomizing arm. Other secondary endpoints such as quality of life or pain intensity will also be assessed blindly from the randomizing arm (patient assessment). Blinding of the surgeon is not possible. The device cannot be blinded from the surgeon's view.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-DYN Device (Experimental): The surgical technique for placement of the B-Dyn device is performed under general anaesthesia. The procedure begins with the insertion of the first upper polyaxial screw which is screwed in with the polyaxial screwdriver. The use of the phantom (Trial 10) is necessary in order to position the second screw. Once the screws are positioned, the B-Dyn is taken between the jaws of the gripping forceps in order to insert it into the heads of the polyaxial screws. The movable rod of the B-Dyn is then placed in the head of the upper screw. The positioning mark of the fixed rod must be placed facing the operator and in the center of the lower screw head. Finally the cap of the lower polyaxial pedicle screw is tightened. A final tightening of the two plugs on the polyaxial pedicle screw heads is performed to fix the assembly.
  Interventions: Device: B-DYN
- Conventional bolted fusion (with or without cage) (Active Comparator): The surgeon will complete his gesture by placing 2 screws in the upper vertebra and 2 screws in the lower vertebra; the screws will be connected to each other to stabilize the assembly. This type of surgery is done via posterior approach and under general anaesthesia.
  Interventions: Device: Conventional Bolted fusion (with or without cage)

INTERVENTIONS:
Device: B-DYN — The surgical technique for placement of the B-Dyn device is performed under general anaesthesia. The procedure begins with the insertion of the first upper polyaxial screw which is screwed in with the polyaxial screwdriver. The use of the phantom (Trial 10) is necessary in order to position the second screw. Once the screws are positioned, the B-Dyn is taken between the jaws of the gripping forceps in order to insert it into the heads of the polyaxial screws. The movable rod of the B-Dyn is then placed in the head of the upper screw. The positioning mark of the fixed rod must be placed facing the operator and in the center of the lower screw head. Finally the cap of the lower polyaxial pedicle screw is tightened. A final tightening of the two plugs on the polyaxial pedicle screw heads is performed to fix the assembly.
  Arms: B-DYN Device
Device: Conventional Bolted fusion (with or without cage) — The surgeon will complete his gesture by placing 2 screws in the upper vertebra and 2 screws in the lower vertebra; the screws will be connected to each other to stabilize the assembly. This type of surgery is done via posterior approach and under general anaesthesia.
  Arms: Conventional bolted fusion (with or without cage)

SUMMARY:
Degenerative Lumbar Spinal Stenosis (LSS) is an extremely common condition affecting more than 102 million people each year. It is a narrowing of the spinal canal in the lower back. It causes pain and even disorders of the lower limbs. When the symptoms get worse and the individual feels functional discomfort despite medical treatment, surgical intervention is recommended. Two surgical options are available: Rigid Stabilization Devices as conventional fusion with or without cage, or dynamic stabilization system as B-DYN device, this system is called "dynamic" because it allows the stabilization of the operated part while preserving a certain mobility.

The main objective of this study is to evaluate the efficacy and tolerance of B-Dyn versus conventional bolted fusion (with or without cage) in the treatment of degenerative lumbar stenosis (DLS) on the degree of postoperative functional incapacity. So the investigator's hypothesis is that the use of the B-DYN device in the treatment of DLS could lead to the maintenance of functional disability related to low back pain (maintenance of walking and mobility).

Another important point to be demonstrated in this study is the preservation of the mobility of the stage overlying the assembly performed by B-Dyn. Indeed, the continued degeneration of segments adjacent to lumbar vertebral fusions is a concern for surgeons For B-Dyn, which is a dynamic stabilization, the combination of rigid and flexible parts allows the mobility of the overlying stage to be preserved and could also lead to a decrease in adjacent syndrome in the long-term compared to the use of conventional fusion.

The duration of patient follow-up is 60 months. The inclusion period is 56 months to recruit the necessary number of subjects for the study (a total of 216 patients is expected).

DETAILED DESCRIPTION:
The Lumbar Spinal Stenosis: LSS is an extremely common pathology that affects more than 102 million people worldwide every year.

It is most often linked to the combination of a disk space narrowing (loss of height and bulging within the canal), a hypertrophy of the yellow ligament and of the joint capsules and also a bone overgrowth by the posterior vertebral joints. This may be associated with Grade I spondylolisthesis.

This pathology often extends over several levels, frequently two (L5S1, L4L5 or L4L5, L3L4) sometimes more. A relatively homogeneous group of patients falls within the group of stenosis, from S1 to L2, without significant deviation (scoliosis or cyphosis type).

A wide variety of different surgical techniques are used to treat patients with LSS and patients who have symptoms despite well-conducted medical treatment. Decompressive laminectomy may prove to be insufficient when several levels are affected and also due to the fears of instability induced by the gesture itself (the joint hypertrophy responsible for nerve root compression is also a stabilizing element). Therefore, the scientific community usually associates a gesture of stabilization with the gesture of decompression.

The choice of stabilizing means is discussed without any conclusive answer provided by any controlled study. This question accounts for the subject of this study.

Two alternatives are discussed:

* The current gold standard is to practice rigid stabilization through bolted fusion, with or without inter somatic cage, despite the fact that it causes an excessive rigidification of the mobile segment, therefore responsible for the acceleration of the degeneration of the upper level.
* Soft stabilization system with pedicular screwing B-Dyn type. It stabilizes the arthrodesis while maintaining some mobility. This partial preservation of mobility could slow down or prevent the upper level's degradation.

Based on the judgment from the dynamic profile images, the devices, some of which are approved in the USA claim to favor fusion while providing no information on the mobility of the upper level in their studies.

The aim of this randomized and prospective comparative study would not only be to establish the non-inferiority of the procedure under study, versus conventional fusion (with or without cage) on the degree of functional disability after surgery, but also to demonstrate the significantly higher preservation of the upper level's mobility when assembling.

First inclusion : May 2020

Inclusion period : 56 months

Follow up of the last patient: December 2029

Analysis and results: June 2030

ELIGIBILITY:
Inclusion Criteria:

Disease related criteria:

1. Stenosis on 1, 2 or 3 disc levels (grade B or C or D according to Schizas classification or central stenosis of grade A according to Schizas classification with a lateral stenosis (postero-lateral overhang or disc protrusion)) on MRI (lumbar spine MRI )
2. Spondylolisthesis grade 1 or no the upper surgical (treated) level
3. Neurological impairment or neurogenic claudication on one or both legs (VAS score > 30)
4. Subjects who have failed well-managed medical treatment that has not resulted in long-lasting symptom relief (duration of symptoms > 3 months);
5. Subjects with no contraindication to fusion or the application of B-Dyn®.

Population-related criteria

1. Subjects of both sexes, 40 years of age and older
2. Subjects who have given free, informed and written consent to participate in the study;
3. Subjects who are able to respond to questionnaires and who can communicate in the language of the study country ;
4. Subjects affiliated to a social security scheme or entitled to a social security scheme.

Exclusion Criteria:

Disease related criteria:

1. Spondylolisthesis of grade > 1 on the upper surgical (treated) level
2. Intervention required on more than 3 disc levels
3. Degenerative Scoliosis (Cobb angle > 20°);
4. Stenosis located only on the L5-S1 level
5. History of instrumented lumbar surgery (cage, rod, etc.) on the upper or lower level, except in the case of instrumentation of the lower level with an intra-spinous device.
6. Stenosis not caused by from degenerative changes.
7. Isolated disc herniation
8. Other specific vertebral damage (for example: ankylosing spondylitis, cancer or neurological disorders)
9. History of vertebral compression fractures at the instrumented level
10. History of osteoporotic fractures
11. Psychological disorders (e.g. dementia ….etc) or drug addiction that lead to an inability to participate in the study
12. Chronic infection

Population related criteria:

1. Withdrawal of consent;
2. Pregnant or Breastfeeding woman
3. Participation in a clinical trial in the 3 months prior to the initial visit;
4. Predicted unavailability during study. Patient deprived of liberty or under guardianship.

Medical Device related criteria:

1. Allergy to any of the components of the medical device.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of change from baseline degree of functional disability, related to low back pain, by using the Oswestry Disability Index (ODI) at 12th month post-surgery | Baseline, 12 months
  The Oswestry questionnaire helps assess the symptoms and severity of back pain, as well as the impairment on daily life activities. The questionnaire contains 10 questions, concerning: pain, personal care, loads, walking ability, sitting position, standing position, sleep, sexual life, social life, travels. Each question offers 6 answers, with a score of 0 to 6 that the patient must choose; score 0 corresponds to a normal function, and score 6 to a very diminished function. The score obtained is multiplied by 2 to get a percentage of disability, with 0% for the absence of disability, and 100% for the most important disability. Completion of the test takes about 5 minutes

SECONDARY OUTCOMES:
Measuring the mobility of the upper instrumented level and adjacent levels at inclusion, 2 months, 12 months and 60 months post intervention using dynamic X-rays of the lumbar spine: | Inclusion, at 2 months, at 12 months and at 60 months
  Dynamic X-ray is a radiograph to measure the mobility of instrumented level and adjacent one. During this radiograph, the patient will be asked to bend down until he/she reaches the painful threshold in flexion and extension, and in lateral inclination. This image should focus on the instrumented level. The degree of mobility is calculated by subtracting the angle that is formed in flexure by the tangent of the upper layer of the upper vertebra, and the tangent of the lower layer to the angle formed by these extending tangents.
Measuring the evolution of the degree of functional disability related to lumbar and radicular pain by the Oswestry Disability Index (ODI) at inclusion, 2 months, 12 months, 24 months and 60 months post-intervention; | Inclusion, at 2 months, at 12 months, 24 months, and at 60 months
  The Oswestry questionnaire helps assess the symptoms and severity of back pain, as well as the impairment on daily life activities. The questionnaire contains 10 questions, concerning: pain, personal care, loads, walking ability, sitting position, standing position, sleep, sexual life, social life, travels. Each question offers 6 answers, with a score of 0 to 6 that the patient must choose; score 0 corresponds to a normal function, and score 6 to a very diminished function. The score obtained is multiplied by 2 to get a percentage of disability, with 0% for the absence of disability, and 100% for the most important disability. Completion of the test takes about 5 minutes
Assessing the intensity of radicular and lumbar pain by the VAS scale (0-100) at inclusion, 2 months, 12 months, 24 months and 60 months post-intervention; | Inclusion, at 2 months, at 12 months, 24 months, and at 60 months
  The visual analogue scale is shaped as a graduated ruler: from 0 to 100; 0 means that the subject has no pain and 100 is the maximum pain he can bear. It's a self-assessment scale. It is sensitive, reproducible, reliable and validated in both acute and chronic pain situations.
Assessing the quality of life by the Short Forum Health Survey(SF-12 score) at inclusion, 2 months, 12 months, 24 months and 60 months post-intervention; | Inclusion, at 2 months, at 12 months, 24 months, and at 60 months
  The Short Forum Health Survey (SF-12 test) is an abbreviated version of the Medical Outcomes Study Short-Form General Health Survey (SF-36) with only 12 of the 36 questions. The SF-12 provides two scores: a mental and social quality of life score and a physical quality of life score. The maximum value is 56 and the minimum value is 12. Higher Scores indicates better physcial and mental health
Measuring the anxiety using the Hospital Anxiety and Depression Scale (HAD) at inclusion, 2 months, 12 months, 24 months and 60 months post-intervention; | Inclusion, at 2 months, at 12 months, 24 months, and at 60 months
  The HAD scale is a tool that detects anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. There are seven questions related to anxiety (total A) and seven others related to the depressive dimension (total D); this provides two scores (maximum score of each score = 21)
Assessing the motion status at the instrumented level and adjacent levels (right and left), by measuring motor skills at inclusion, 2 months, 12 months and 60 months post-intervention | Inclusion, at 2 months, at 12 months and at 60 months
  MRC scale will be used to evaluate the motor function: 0 means no movement/contractions, 5 means normal muscle strength). The neurological status will be assessed at the L4, L5 and S1 levels (right and left)
Assessing the sensory status at the instrumented level and adjacent levels (right and left), by measuring feeling of touch and stinging sensation at inclusion, 2 months, 12 months and 60 months post-intervention | Inclusion, at 2 months, at 12 months and at 60 months
  MRC scale for sensory assesment will be used to assess the sensation of touch and sting : 0 means Absent and 2 means Normal. The motor status will be assessed at the L4, L5 and S1 levels (right and left)
Measuring different radiological parameters as lumbar lordosis (LL), instrumented level segmental lordosis, disk height, pelvic parameters by full spine radiograph | Inclusion, at 2 months, at 12 months and at 60 months
  Full spine radiograph (EOS) is a face and profil X-ray, on which the sagittal alignment parameters will be measured. An independent radiologist will be in charge of the centralized reading.
Evaluation of the maximum walking distance by self-paced test | Inclusion, at 2 months, at 12 months and at 60 months
  Self-Paced Walking Test (SPWT) assesses walking capacity by measuring the total distance the patient can continuously walk on a flat surface at a self-selected pace, until experiencing symptoms of LSS or reaching a limit of 30 minutes.
The rate of re-intervention on the instrumented level or adjacent level during the study | During the whole study (up to 60 months)
  A re-operation during the study is defined as a secondary intervention at the instrumented level or adjacent level for any reason (infectious or mechanical): revision, implant removal (explantation), fusion, need for additional fixation. etc
Evaluation of radiological adjacent syndrome by simple and dynamic radiology and MRI. | 60 months
  Radiological adjacent syndrome is considered if in simple and dynamic radiology, we will detect the narrowing of the disc height (> 3 mm), posterior opening ( > 5°) and sliding progression (> 3 mm) compared to the pre-operative data of the lateral bending radiology.
  Using MRI, we will follow postoperation progression of disc degeneration according to the Pfirrmann classification and the progression of spinal canal stenosis according to the classification of Imagama.
  The 1 grade progression of disk degeneration or spinal canal stenosis on MRI is considered an adjacent radiological syndrome.
Evaluation of symptomatic adjacent syndrome adjacent syndrome | 60 months
  Symptomatic adjacent syndrome is considered when clinical symptoms such as radicular pain of the segment adjacent to the treated level is confirmed by using the visual analogue scale (shaped as a graduated ruler: from 0 to 100; 0 means that the subject has no pain and 100 is the maximum pain he can bear) .
Evaluation of surgical adjacent syndrome | 60 months
  Surgical adjacent syndrome is considered if additional operation to treat clinical symptoms such as radicular pain (assessed using the visual analogue scale graduated from 0 to 100; 0 means that the subject has no pain and 100 is the maximum pain he can bear) of the segment adjacent to the treated level is required.
Assessing safety and tolerance | During the whole study (up to 60 months)
  By evaluating Number of patients who experienced at least one adverse event during the follow-up period.
Assessing safety and tolerance | During the whole study (up to 60 months)
  By evaluating Number of patients who experienced a serious adverse event during the follow-up period.
Assessing safety and tolerance | During the whole study (up to 60 months)
  By evaluating Rate of short and long-term intraoperative and post-operative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent POINTILLART, Professor, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU [University Hospital Center]of Bordeaux - Le Tripode - GH Pellegrin/ Department of Orthopaedic and Trauma Surgery Spinal Surgery Unit, Bordeaux
  - Clinique Des Cedres, Cornebarrieu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravindra VM, Senglaub SS, Rattani A, Dewan MC, Hartl R, Bisson E, Park KB, Shrime MG. Degenerative Lumbar Spine Disease: Estimating Global Incidence and Worldwide Volume. Global Spine J. 2018 Dec;8(8):784-794. doi: 10.1177/2192568218770769. Epub 2018 Apr 24. PMID 30560029
- [Background] Turner JA, Ersek M, Herron L, Deyo R. Surgery for lumbar spinal stenosis. Attempted meta-analysis of the literature. Spine (Phila Pa 1976). 1992 Jan;17(1):1-8. doi: 10.1097/00007632-199201000-00001. PMID 1531550
- [Background] Machado GC, Ferreira PH, Yoo RI, Harris IA, Pinheiro MB, Koes BW, van Tulder MW, Rzewuska M, Maher CG, Ferreira ML. Surgical options for lumbar spinal stenosis. Cochrane Database Syst Rev. 2016 Nov 1;11(11):CD012421. doi: 10.1002/14651858.CD012421. PMID 27801521
- [Background] Radcliff KE, Kepler CK, Jakoi A, Sidhu GS, Rihn J, Vaccaro AR, Albert TJ, Hilibrand AS. Adjacent segment disease in the lumbar spine following different treatment interventions. Spine J. 2013 Oct;13(10):1339-49. doi: 10.1016/j.spinee.2013.03.020. Epub 2013 Jun 15. PMID 23773433
- [Background] Morishita Y, Ohta H, Naito M, Matsumoto Y, Huang G, Tatsumi M, Takemitsu Y, Kida H. Kinematic evaluation of the adjacent segments after lumbar instrumented surgery: a comparison between rigid fusion and dynamic non-fusion stabilization. Eur Spine J. 2011 Sep;20(9):1480-5. doi: 10.1007/s00586-011-1701-1. Epub 2011 Feb 8. PMID 21301893

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT04407338/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT04407338/ICF_001.pdf